CLINICAL TRIAL: NCT00004751
Title: Phase II Randomized Study of Selective Dorsal Rhizotomy and Physiotherapy Vs Physiotherapy Alone for Spastic Diplegia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Collaborators: Seattle Children's Hospital (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 199/11667; CHS-01699211
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1997-02

CONDITIONS: Spastic Diplegia
Keywords: cerebral palsy; neurologic and psychiatric disorders; rare disease; spastic diplegia
MeSH Terms: conditions — Cerebral Palsy; Neurologic Manifestations; Mental Disorders; Rare Diseases | interventions — Surgical Procedures, Operative; Physical Therapy Modalities

INTERVENTIONS:
Procedure: Surgery
Procedure: Physical therapy

SUMMARY:
OBJECTIVES:

I. Assess the efficacy and safety of selective dorsal rhizotomy and physiotherapy compared with physiotherapy alone in improving gross motor function and reducing spasticity in children with spastic diplegia.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized study. Patients are stratified by age and the ability to ambulate 50 feet unaided. Each stratum is block randomized.

Patients are randomly assigned to surgery plus intensive physical therapy versus intensive physical therapy alone.

The surgical procedure is a selective dorsal rhizotomy. Physical therapy (PT) includes passive and active range of motion, facilitation of isolated muscle control, transitional movements, strengthening, transfer skills, and gait training. The PT schedule is 2-hour sessions 5 days a week for 1 month, 1-hour sessions 5 days a week for 5 months, then a standard therapy program for the remainder of the study (total of 6 months). Parents supervise exercise on non-PT days.

Patients are followed at 6, 12, and 24 months.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Spastic diplegia, i.e.: Measurable spasticity with more lower than upper limb involvement
* Fair to good trunk and head control
* Little or no bulbar involvement
* Able to walk or has potential to walk indoors with assistive devices
* No fixed musculoskeletal deformity greater than 15 degrees
* Prior orthopedic surgery acceptable if spastic muscle group is in physiologic biomechanical position and retains voluntary power
* No detectable athetosis, rigidity, ataxia, or other movement disorder
* No disease-related, treatable condition that may become urgent during study, e.g., hip subluxation requiring adductor release

--Patient Characteristics--

* Age: 3 to 18
* Other: Intelligence Quotient greater than 50 Developmental age 3 years or higher
* Able to follow multi-step commands
* Expressive communication skills at 3-year level or higher
* Mild dysarthria or drooling does not exclude
* Stable social environment
* Regular school and physical therapy attendance
* Normal psychiatric status
* Guardian able to give support and follow-up care
* No medical contraindication to anesthesia or surgery, e.g.: Previous anesthesia reaction
* Chronic lung disease
* Uncontrollable seizures
* Scoliosis Vertebral anomaly
* Neural tube defect
* No visual impairment sufficient to hinder mobility
* Able to come to Children's Hospital and Medical Center for follow-up Insurance coverage adequate for surgery and postoperative physiotherapy

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 1991-10

CONTACTS AND LOCATIONS:
Overall Officials: John F. McLaughlin, Study Chair — Seattle Children's Hospital